CLINICAL TRIAL: NCT02423499
Title: Features Emotional Responses in Adults With Autism: Comparison With Bipolar Disorder
Brief Title: Features Emotional Responses in Adults With Autism: Comparison With Bipolar Disorder (REMBAU)
Acronym: REMBAU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHAO13-ML/REMBAU; 2014-A00431-46 (Other: EudraCT number)
Record Dates: First submitted 2015-04-03; First posted 2015-04-22 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorder; Bipolar Disorder
Keywords: Autism Spectrum Disorder; Bipolar Disorder; Emotions
MeSH Terms: conditions — Autism Spectrum Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autism Spectrum Disorder: Autism Spectrum Disorder adults without intellectual disability
- Bipolar Disorder: Bipolar Disorder adults during normothymic phase of illness
- Healthy Volonteers: Healthy adults

SUMMARY:
The objective of this study is to identify the specific characteristics of Autism Spectrum Disorder (ASD) in emotional response profiles and shared with Bipolar Disorder (BD) characteristics.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  * Age between 18 and 50 years
  * Normal vision (or corrected)
  * Absence of neurological disorder (epilepsy , head trauma, ... )
  * Ability to understand information about the protocol
  * Informed and signed consent
  * normal mood (euthymia)
  * normal or high intelligence
* Subjects with ASD:

  * Subjects with an autism spectrum disorder according to the DSM-5
  * The diagnosis is confirmed by diagnostic interviews: ADI- R (Autism Diagnostic Interview-Revised) and / or ADOS (Autism Diagnostic Observation Schedule ) .
* Subjects with bipolar disorder:

  * Diagnosis of bipolar disorder according to DSM-IV-TR or DSM -5
  * The diagnosis is confirmed by the MINI 6.0 (The Mini-International Neuropsychiatric Interview) .
* Healthy volunteers:

  * Inclusion after checking the national register of healthy volunteers
  * No history of disease of the central nervous system or psychiatric disorder
  * No family history of ASD or BD in the first degree
  * Lack of psychotropic medication or current cardiotropic
  * Lack of psychiatric disorder on Axis I MINI 6.0
  * AQ Score < 32

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ASD subjects will be recruited at Centre Universitaire de Pédopsychiatrie, CHRU de Tours, FRANCE.
  BD subjects will be recruited at Clinique Psychiatrique Universitaire, CHRU de Tours, FRANCE.
  Healthy volunteers will be recruited at Centre d'Inverstigation Clinique, CHRU de Tours, FRANCE.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-05-19 (Actual); Primary Completion 2021-05-26 (Estimated); Study Completion 2021-05-26 (Estimated)

PRIMARY OUTCOMES:
Physiological emotional response during emotion elicitation in a laboratory session (Pupil size measured by eye tracking, heart rate, electrodermal response, breath rate) during emotion elicitation in a laboratory session | average 1 hour

SECONDARY OUTCOMES:
Subjective emotional response during emotion elicitation in a laboratory session | average 1 hour
Facial emotional response during emotion elicitation in a laboratory session | average 1 hour
Experience sampling method in real life during a week (emotions, activities, social context, burden) | within the first 7 days after inclusion
Physiological emotional response in real life (heart rate, electrodermal response, breath rate, actimetry) | within the first 24h approx. after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique BONNET- BRILHAULT, Pr, Principal Investigator — University Center of Child and Adolescent Psychiatry, University Hospital of Tours; Wissam EL-HAGE, Pr, Principal Investigator — University Psychiatric Clinic, University Hospital of Tours; Valérie GISSOT, MD-PHD, Principal Investigator — Clinical Investigation Center, INSERM 14 15, University Hospital of Tours; Mathieu LEMAIRE, MD-PHD, Study Director — University Center of Child and Adolescent Psychiatry, University Hospital of Tours
Locations (1):
- LEMAIRE, Tours, France